CLINICAL TRIAL: NCT05087940
Title: Treatment of Resistant Hypertension: Cohort Study
Acronym: TRYCORT
Status: Completed | Type: Observational
Sponsor: Galenika AD Beograd (Industry)
Collaborators: Medicinsko društvo za racionalnu terapiju Republike Srbije (MEDRAT) (Unknown)
Responsible Party: Principal Investigator, Slobodan Jankovic, Professor, Galenika AD Beograd
Other Study IDs: TRYCORT 1.1
Record Dates: First submitted 2021-10-12; First posted 2021-10-21 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Resistant Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Resistant hypertension: The adult patients with resistant hypertension which is defined as casual blood pressure during clinical examination of more than 140/90 mmHg despite treatment with optimal or best-tolerated doses of three or more drugs, which should include a diuretic, typically an angiotensin converting enzyme (ACE) inhibitor or an angiotensin receptor blocker (ARB), and a calcium channel blocker (CCB). All reference blood pressures will be taken as a mean of the 2nd and 3rd measurements in physician's office during a single examination, measured at least 3 min apart. The following add-on therapy is available in Serbia, where the study is conducted: an aldosterone receptor blocker (e.g. spironolactone), a loop diuretic (e.g. furosemide), a thiazide in large daily dose, an alpha 1 selective blocker and a beta 1 selective blocker.
  Interventions: Drug: Add-on therapy

INTERVENTIONS:
Drug: Add-on therapy — Add-on drugs prescribed by internal medicine specialists within the routine health care and independently from the study investigators - one of the following: an aldosterone receptor blocker, a loop diuretic, a thiazide in large daily dose, an alpha 1 selective blocker or a beta 1 selective blocker
  Other Names: An aldosterone receptor blocker, or a loop diuretic, or a thiazide in large daily dose, or an alpha 1 selective blocker, or a beta 1 selective blocker

SUMMARY:
This is a multicenter, prospective observational cohort study. It will compare effectiveness and safety of various add-on treatment options in regard to arterial blood pressure control in adult patients with treatment resistant hypertension: an aldosterone receptor blocker (e.g. spironolactone), a loop diuretic, a thiazide in large daily dose, an alpha 1 selective blocker or a beta 1 selective blocker. The add-on therapy will be prescribed to the patients within the scope of their routine medical care, independently from the study investigators. The patients will be followed up for 6 months, with monthly visits and continuous home blood pressure diary kept by the patients themselves.

DETAILED DESCRIPTION:
This is a multicenter, prospective observational cohort study. It will compare effectiveness and safety of various add-on treatment options in regard to arterial blood pressure control in adult patients with treatment resistant hypertension: an aldosterone receptor blocker (e.g. spironolactone), a loop diuretic, a thiazide in large daily dose, an alpha 1 selective blocker or a beta 1 selective blocker. The add-on therapy will be prescribed to the patients within the scope of their routine medical care, independently from the study investigators. Both office and home blood pressure measures will be recorded at baseline and then every month for 6 visits. The systolic and diastolic blood pressure targets are chosen according to European guidelines for treatment of hypertension, i.e. < 140/90 mmHg. Participants will have contact with the study team at any time to obtain information on interim study outcomes (updated medical history, completion of study questionnaires). Before, during and after the study the patients will be cared for by their chosen general practitioners independently from the study investigators and referred to internal medicine specialists as necessary, according to diagnostic and treatment protocols currently in power at the study sites. Role of the study investigators will be limited to observation and collection of data from the patients themselves and from their medical files.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Resistant hypertension is defined as casual blood pressure during clinical examination of more than 140/90 mmHg despite treatment with optimal or best-tolerated doses of three or more drugs, which should include a diuretic, typically an angiotensin converting enzyme (ACE) inhibitor or an angiotensin receptor blocker (ARB), and a calcium channel blocker (CCB) (or beta blocker). All reference blood pressures will be taken as a mean of the 2nd and 3rd measurements in physician's office during a single examination, measured at least 3 min apart
3. Aged 18 years or above
4. Inadequate control of hypertension is confirmed with home blood pressure monitoring (average of morning and evening measurements after 5 minutes of relaxation in sitting position, for 6 days)

Exclusion Criteria:

1. Pregnancy, anticipated pregnancy, or breastfeeding
2. Incarceration or institutionalized living which may prohibit measurement of home blood pressure
3. Participation in another intervention study that may affect blood pressure
4. Patients in whom systolic blood pressure is not measurable (e.g. those with left ventricular assist devices)
5. Hypotension: average systolic blood pressure <100 mmHg over last 2 weeks prior to screening while not taking any blood pressure medications
6. Life expectancy <4 months
7. Anticipated living donor kidney transplant within 4 months
8. Patients with a systolic blood pressure value over 220 mmHg requiring immediate adjustments of therapy
9. Patients with moderate to severe renal insufficiency (acute or chronic) with glomerular filtration rate of less than 30 ml/min
10. Patients with active bronchospastic disorders
11. Heart failure classes III and IV
12. Severe bradycardia (heart rate below 50/min), 2nd and 3rd degree AV block
13. Patients with a history of hypersensitivity to any of the drugs under study
14. Patients already using add-on therapy

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects with resistant hypertension (casual blood pressure during clinical examination of more than 140/90 mmHg despite treatment with optimal or best-tolerated doses of three or more drugs, which should include a diuretic, typically an angiotensin converting enzyme (ACE) inhibitor or an angiotensin receptor blocker (ARB), and a calcium channel blocker (CCB) who meet the inclusion and exclusion criteria will be eligible for participation in this study.
Sampling Method: Non-Probability Sample
Enrollment: 731 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Rate of normalization of arterial blood pressure | 6 months
  Decrease of arterial blood pressure to normal levels according to the 2018 European Society for Cardiology (ESC)/European Society for Hypertension (ESH) Guidelines (<140/90 mmHg) after 1,2,3,4,5 and 6 months
Rate of reduction of systolic arterial blood pressure | 6 months
  Reduction of systolic arterial blood pressure for 10 mmHg or more after 1,2,3,4,5 and 6 months
Rate of reduction of diastolic arterial blood pressure | 6 months
  Reduction of diastolic arterial blood pressure for 5 mmHg or more after 1,2,3,4,5 and 6 months
Adverse events rate | 6 months
  Incidence of adverse events
Treatment withdrawal rate | 6 months
  Tolerability

SECONDARY OUTCOMES:
Blood pressure | 6 months
  Absolute value of arterial blood pressure at scheduled study visits
Renal function | 6 months
  Parameters of renal function - serum level of creatinine and absolute value of proteinuria
Quality of life on a scale 0 to 1 | 6 months
  Quality of life at a visual analogue scale

CONTACTS AND LOCATIONS:
Overall Officials: Branko Andjelkovic, MD, Study Director — GALENIKA; Slobodan Jankovic, DSc, MD, Principal Investigator — University of Kragujevac, Faculty of Medical Sciences
Locations (12):
- Serbia (12):
  - Clinical Center of Serbia, Belgrade
  - Clinical Hospital Center Zemun, Belgrade
  - Clinical Hospital Center Zvezdara, Belgrade
  - Medical Military Academy, Belgrade
  - University Clinical Hospital Center Dragisa Misovic - site 1, Belgrade
  - University Clinical Hospital Center Dragisa Misovic - site 2, Belgrade
  - University Hospital Medical Center Bezanijska Kosa, Belgrade
  - Institute of Cardiovascular Diseases of Vojvodina, Kamenitz
  - University Clinical Center Kragujevac, Kragujevac
  - General Hospital Leskovac, Leskovac
  - Clinical Center Nis, Niš
  - General Hospital Subotica, Subotica

IPD SHARING:
Plan to Share IPD: No